CLINICAL TRIAL: NCT06702696
Title: Consumption of Anti-Inflammatory Effects of Aronia (Aronia Melanocarpa) Berry in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Aronia Berry Consumption on Inflammatory Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Buse Sarıkaya, Principal Investigator Research Assistant Dr. Buse Sarıkaya, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SarikayaB.
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: anti-inflammatory; black chokeberry; COPD; aronia melanocarpa; cytokines
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aronia group (Experimental): The Aronia group will consume 30 g of freeze-dried aronia powder (n=25).
  Interventions: Dietary Supplement: Black chokeberry (Aronia melanocarpa)
- Placebo group (Placebo Comparator): The placebo group will consume placebo powder (n=25).
  Interventions: Other: Placebo powder

INTERVENTIONS:
Dietary Supplement: Black chokeberry (Aronia melanocarpa) — The aronia group, who will consume 30 g of freeze-dried aronia powder (n=25)
  Arms: Aronia group
Other: Placebo powder — The placebo group, who will consume placebo powder (n=25).
  Arms: Placebo group

SUMMARY:
The study will aim to evaluate the effects of consuming freeze-dried aronia berries as an adjunct to medical treatment in patients with chronic obstructive pulmonary disease (COPD), focusing on anti-inflammatory, respiratory, and biochemical parameters.

It will be conducted at a research hospital in Istanbul, involving 50 participants aged 50-80 diagnosed with COPD. Participants will be randomly assigned to two groups: the aronia group (AG, n=25) and the placebo group (PG, n=25). The AG will receive 30 g of freeze-dried aronia powder daily, while the PG will receive 30 g of placebo powder, both for a duration of 8 weeks. Baseline demographic data will be collected through face-to-face interviews, while biochemical, respiratory, anthropometric, and body composition parameters will be assessed both before and after the intervention. Dietary intake records will also be collected and analyzed.

DETAILED DESCRIPTION:
Participant Selection This study will be conducted between November 15, 2024, and November 15, 2025, at the Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital Pulmonology Outpatient Clinic. Participants will include patients who will be diagnosed with COPD by a physician. The diagnosis of COPD will be based on spirometry, specifically when Forced Expiratory Volume in 1 second): FEV1 is below 80% of the predicted value.

COPD cases will be classified according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2020 Guidelines. Post-bronchodilator FEV1 values will categorize patients into mild (FEV1 ≥ 80% predicted), moderate (50% ≤ FEV1 < 80% predicted), severe (30% ≤ FEV1 < 50% predicted), or very severe (FEV1 < 30% predicted). Sample size calculations will assume a detectable change of 0.67 pg/mL in the primary outcome variable (Tumor Necrosis Factor-alpha, TNF-α) at a significance level of 0.05 and a power of 0.80. These calculations will be performed using the software available at http://hedwig.mgh.harvard.edu/sample_size/js/js_crossover_quant.html.

Acquisition and Preparation of Aronia Berries Aronia berries (Aronia melanocarpa) will be obtained in season from the Atatürk Horticultural Central Research Institute of the Turkish Ministry of Agriculture and Forestry. The berries will be freeze-dried using a TRS-2-4 lyophilizer at -55°C. A single fruit exchange (containing 15 g of carbohydrates) will correspond to 200 g of lyophilized aronia berries, which will be vacuum-packed for participant use.

Study Design This study will be designed as a randomized, placebo-controlled, double-blind trial. Patients diagnosed with COPD at the Yedikule Pulmonology Clinic and willing to volunteer will be included after providing informed consent. Fifty participants (25 male, 25 female) who meet the study criteria will be randomized into two groups using a sealed envelope method.

The placebo will consist of maltodextrin combined with oil-based berry flavoring, citric acid, powdered sugar, pink-black food coloring, and liquid oil as a solvent for the flavoring. Placebos will be provided in 30 g vacuum-sealed packets and will be indistinguishable from the aronia supplements in color and weight.

The intervention phase will last eight weeks. Physicians, researchers, and participants will remain blinded to the type of product consumed (aronia or placebo). Participants will record their dietary intake during the study, and a food diary will be collected for nutritional assessment. Clinical evaluations will occur twice: at baseline and at the end of the 8th week following randomization.

Data Collection and Assessment Data will be collected using a questionnaire developed by the researchers based on literature reviews, administered via face-to-face interviews. The questionnaire will include 20 questions covering demographics, health status, physical activity, dietary habits, weight changes, and appetite loss over the past six months. Participants will also complete a COPD Assessment Test (CAT) and record food intake. Anthropometric measurements, spirometry, and biochemical tests will be conducted, and blood samples will be collected for analysis.

To minimize daily variations, all assessments will be conducted between 8:00 and 10:00 AM, following an overnight fast (after 10:00 PM the previous night). At baseline, participants will complete a demographic survey during face-to-face interviews, and all participants will sign a written informed consent form.

Dietary Intake Records Participants' dietary intake will be evaluated before and after the intervention using a one-day food record. The food records will be obtained through face-to-face interviews and will include meal components, preparation methods, quantities, measurements, and, for processed or enteral products, brand names. Nutritional assessments will be performed using the BeBis 9.0 software, and results will be compared with the Turkey Dietary Guidelines (TÜBER) to calculate the percentage of daily nutrient requirements met. Intakes below 50% of daily recommendations will be considered insufficient.

Body Composition and Anthropometric Measurements Body composition will be assessed using bioelectrical impedance analysis (BIA) with an eight-electrode InBody 120 device (InBody Co., Ltd., Istanbul, Turkey). Measurements will be conducted after a minimum of 8 hours of fasting, with participants barefoot and standing in an upright position. Parameters measured will include body weight (kg), skeletal muscle mass (kg), body fat mass (kg), body fat percentage (%), total body water (L), and visceral fat level.

Anthropometric measurements will include height (m), waist circumference (cm), and mid arm circumference. Height will be measured with a portable InBody stadiometer in a standing position without shoes. Waist circumference will be measured at the midpoint between the lowest rib and the iliac crest, while mid arm circumference will be taken from the non-dominant arm at the midpoint between the acromion and olecranon.

Spirometry Lung function tests will be performed by trained spirometry technicians at the hospital. Patients will take three normal breaths, then perform a maximum inhalation followed by a forceful exhalation to measure Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), and the FEV1/FVC ratio.

The FEV1 refers to the volume of air exhaled in the first second of the forced breath. The FVC represents the total volume of air forcibly exhaled after a full inhalation. The FEV1/FVC ratio, expressed as a percentage, indicates the proportion of the FVC exhaled during the first second, serving as a key parameter for assessing airflow obstruction.

COPD Assessment Test (CAT) The CAT will evaluate the impact of COPD on patients' lives, including symptoms such as cough, sputum, breathlessness, fatigue, and confidence in leaving home. Validity and reliability for Turkish patients were established by Yorgancıoğlu et al. The CAT is an eight-item, self-administered questionnaire, each item is scored on a scale of 0 to 5, resulting in a total score ranging from 0 to 40, with higher scores indicating greater health impairment.

Biochemical Analyses Blood samples (5 mL) will be collected from fasting participants, centrifuged at 3000 g for 10 minutes, and stored in serum separator tubes. Serum samples will be preserved using a cold chain for biochemical analysis. Further details regarding the analyses will be available in the study protocol

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-80 years
* Diagnosed with COPD
* Not following a vegetarian or vegan diet
* Willing to consume the provided aronia berry (black chokeberry)
* Non-smokers
* Have signed the informed consent form
* Has not undergone endobronchial tube or valve surgery in the last two years.

Exclusion Criteria:

* Presence of associated chronic inflammatory/rheumatic diseases
* Chronic infections that may create a prothrombotic state
* Chronic kidney disease (CKD)
* Malignancy
* Hereditary thrombophilia
* Essential thrombocythemia
* Diagnosed endocrine disorders
* Malabsorption disorders
* Allergy to any food or berry fruits
* Smoking
* Participants who did not sign the informed consent form

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein (CRP) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Serum CRP levels will be measured to evaluate systemic inflammation in participants. The results will be reported in picograms per milliliter (pg/mL).
Tumor Necrosis Factor-Alpha (TNF-Alpha) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Serum TNF-alpha levels will be analyzed as a marker of inflammation. The results will be reported in nanograms per liter (ng/L).
Interleukin-1 Beta (IL-1β) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Serum IL-1β levels in serum will be measured as an indicator of pro-inflammatory activity. Results will be reported in picograms per milliliter (pg/mL).
Interleukin-6 (IL-6) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Serum IL-6 levels will be assessed as a biomarker of inflammation. The measurements will be conducted using enzyme-linked immunosorbent assay (ELISA) and reported in nanograms per liter (ng/L).
Interleukin-8 (IL-8) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Serum IL-8 levels will be assessed as a biomarker of inflammation. The measurements will be conducted using enzyme-linked immunosorbent assay (ELISA) and reported in nanograms per liter (ng/L).
Interleukin-10 (IL-10) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Serum IL-10 levels will be assessed as a biomarker of inflammation. The measurements will be conducted using enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Total Antioxidant Status (TAS) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  TAS will be measured spectrophotometrically to evaluate the total antioxidant capacity in serum. Results will be expressed as millimoles per liter ascorbate equivalent (mmol/L Ascorbate Eq). TAS and Total Oxidant Status (TOS) will be combined to report Oxidative Stress Index (OSI).
Total Oxidant Status (TOS) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  TOS will be analyzed spectrophotometrically to assess the overall oxidative stress in serum. Results will be expressed as micromoles of hydrogen peroxide equivalent per liter (µmol H2O2 Eq/L). TAS and TOS will be combined to report Oxidative Stress Index (OSI).
The Oxidative Stress Index (OSI) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  (OSI) is calculated as the ratio of TOS to TAS. This ratio represents the balance between oxidants and antioxidants in a system. Result will be expressed as an arbitrary unit (AU).
COPD Assessment Test (CAT) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  The COPD Assessment Test will be used to evaluate the health status of participants with COPD. The CAT score will range from 0 to 40, with higher scores indicating greater health impairment.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  FVC will be assessed using spirometry and reported in liters (L). The assessment will measure the maximum volume of air a participant can forcibly exhale after a full inhalation. FVC and Forced Expiratory Volume in 1 Second (FEV1) will combined to report FVC/FEV1 ratio.
Forced Expiratory Volume in 1 Second (FEV1) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  FEV1 will be measured using spirometry and reported in liters (L). The test evaluates the volume of air exhaled in the first second of a forceful exhalation. FVC and FEV1 will combined to report FVC/FEV1 ratio.
FVC/FEV1 Ratio | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  The ratio of forced vital capacity (FVC) to forced expiratory volume in 1 second (FEV1) will be calculated to assess airflow limitation. Results will be expressed as a percentage.

OTHER OUTCOMES:
Fasting Blood Glucose | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Fasting blood glucose levels will be measured to assess participants' glycemic control. Results will be reported in milligrams per deciliter (mg/dL) and reflect glucose concentration after an overnight fast.
Triglycerides (TG) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Triglyceride levels will be measured to assess lipid metabolism. Results will be expressed in milligrams per deciliter (mg/dL).
High-Density Lipoprotein (HDL) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  HDL cholesterol levels will be measured to evaluate cardiovascular risk. Results will be reported in milligrams per deciliter (mg/dL).
Low-Density Lipoprotein (LDL) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  LDL cholesterol levels will be assessed to understand lipid-related cardiovascular risk. Results will be expressed in milligrams per deciliter (mg/dL).
Total Cholesterol | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Total cholesterol levels will be measured to evaluate overall lipid profiles. Results will be reported in milligrams per deciliter (mg/dL).
Weight | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Weight will be measured in kilograms (kg) using a digital scale to assess the participant's overall body weight. Weight and height will be combined to report BMI in kg/m2.
Height | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Height will be measured in centimeters (cm) using a clinical stadiometer to assess participants' stature. Weight and height will be combined to report BMI in kg/m2.
Body Mass Index (BMI) | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  BMI will be calculated using the formula: weight (kg) divided by the square of height (m²). It is used to assess body weight relative to height.
Waist Circumference | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Waist circumference will be measured in centimeters (cm) at the midpoint between the lowest rib and the iliac crest to evaluate abdominal fat distribution with an atropometric measuring tape.
Hip Circumference | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Hip circumference will be measured in centimeters (cm) at the widest point around the hips, using an anthropometric measuring tape, providing an indication of overall fat distribution .
Mid-arm Circumference | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Mid-arm circumference will be measured in centimeters (cm) at the midpoint between the acromion process and the olecranon process of the upper arm to assess upper body mass, using an anthropometric measuring tape.
Skeletal Body Mass | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Skeletal body mass, measured in kilograms (kg), will be assessed using bioelectrical impedance analysis (BIA) to estimate the weight of bones and related structures.
Body Fat Mass | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Body fat mass, measured in kilograms (kg), will be assessed using BIA to estimate the total fat mass in the body.
Body Fat Content | Baseline (T0, 1 week before the beginning of the study); T1 (8 weeks after the end of the treatment/control period).
  Body fat content will be expressed as a percentage of total body weight, indicating the proportion of body weight that is made up of fat. This will be assessed using BIA.

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Göğüs Hastalıkları Hastanesi, Istanbul, Zeytinburnu, Turkey (Türkiye)